CLINICAL TRIAL: NCT04399031
Title: Effects of e-Cigarettes on Perceptions and Behavior - Substudy 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS-18-00839 Substudy 1
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Electronic Cigarette Use; Cigarette Use, Electronic; Vaping; Cigarette Smoking
MeSH Terms: conditions — Vaping; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- E-cigarette e-liquid 1 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 2 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 3 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 4 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 5 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 6 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 7 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 8 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 9 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 10 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 11 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 12 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 13 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 14 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 15 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 16 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 17 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 18 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 19 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid
- E-cigarette e-liquid 20 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Drug: E-cigarette e-liquid

INTERVENTIONS:
Drug: E-cigarette e-liquid — Participants will self-administer an experimenter-provided e-cigarette.

SUMMARY:
This project will assess the ways in which e-cigarette product diversity impacts the user experience to inform potential regulations by identifying product characteristics that may: (1) put young adults at risk for tobacco product use; and (2) facilitate adult smokers switching to e-cigarettes. There are three primary objectives to the study: (1) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect product appeal across young adult e-cigarette users and middle-age/older adult smokers; (2) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect abuse liability in young adult e-cigarette users and the ability to resist smoking in adult smokers; (3) Determine the affect of product characteristics on e-cigarette nicotine delivery profile. For this substudy, young adult vapers (N=100) and adult smokers (N=100) will attend one laboratory session in which they will self-administer e-cigarette products varied according to within-subject e-cigarette factors (e.g., flavor, nicotine formulation).

ELIGIBILITY:
Inclusion Criteria:

Vapers/E-cigarette Users

* E-cigarette/vaping device use at least three days per week for at least 2 months
* Regular use of e-cigarettes/vaping devices containing nicotine

Cigarette Smokers

* Daily cigarette smoking for at least two years
* Currently smoke at least four cigarettes per day
* Interested in trying an e-cigarette or current use of an e-cigarette

Exclusion Criteria:

Vapers/E-cigarette Users

* Pregnant or breastfeeding
* Desire to cut down on use of e-cigarette/vaping device

Cigarette Smokers

* Pregnant or breastfeeding
* Current daily use of other combustible tobacco products (such as cigars)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Subjective Appeal | 1 hour
  Self-report measures of product appeal will be completed following e-cigarette self-administration.
Sensory Appeal | 1 hour
  Self-report measures of product appeal will be completed following e-cigarette self-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Leventhal, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tackett AP, Dai HD, Han DH, Vogel EA, Coreas SI, Jafarzadeh N, Gonzalez Anaya MJ, Patel D, Peraza N, Mason TB, Leventhal AM. Appeal of e-cigarette flavors: Differences between never and ever use of combustible cigarettes. Drug Alcohol Depend. 2023 May 1;246:109849. doi: 10.1016/j.drugalcdep.2023.109849. Epub 2023 Mar 23. PMID 37028103
- [Derived] Leventhal AM, Madden DR, Peraza N, Schiff SJ, Lebovitz L, Whitted L, Barrington-Trimis J, Mason TB, Anderson MK, Tackett AP. Effect of Exposure to e-Cigarettes With Salt vs Free-Base Nicotine on the Appeal and Sensory Experience of Vaping: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2032757. doi: 10.1001/jamanetworkopen.2020.32757. PMID 33433597